CLINICAL TRIAL: NCT04819867
Title: Comparison Of The Effect Of Propolis And Gluma Desensitizer On The Management Of Dentin Hypersensitivity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Marina Shah, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MShah
Record Dates: First submitted 2021-03-12; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Propolis; gluma desensitizer; Gluma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propolis (Experimental): propolis will be applied to the affected teeth
  Interventions: Drug: Propolis
- gluma desensitizer (Active Comparator): Gluma desensitizer will be applied to the affected teeth
  Interventions: Drug: Gluma Desensitizer

INTERVENTIONS:
Drug: Propolis — propolis is an extract derived from bee hives
  Arms: propolis
Drug: Gluma Desensitizer — Gluma is a desensitizer agent
  Other Names: gluma
  Arms: gluma desensitizer

SUMMARY:
Objective The purpose of this study was to compare the effect of Propolis and Gluma desensitizer on the management of Dentin Hypersensitivity Methods Patients with dentin hypersensitivity exhibiting pain scores of at least '2' on the visual analog scale (VAS) were included in the study. Patient's response to an air blast stimulus was noted on Visual Analogue Scale and Schiff's scale in order to record the degree of hypersensitivity of teeth. There were 80 teeth, 40 in each group. The baseline scores were obtained. Propolis and Gluma desensitizer were randomly applied to each hypersensitive tooth. VAS scores and Schiff's sensitivity score for air blast stimulus were then noted at baseline, immediate, after 1 week and then after 1 month of application.

DETAILED DESCRIPTION:
INTRODUCTION Dentin hypersensitivity is commonly characterized by a short sharp pain. This pain is believed to arise from the dentinal tubules that are exposed particularly in response to external stimuli such as evaporative, thermal, tactile or chemical forces.Pain caused by dentin hypersensitivity hampers an individual's day to day activities which includes eating, drinking and often breathing. Since patients do not perceive this as a severe problem they usually do not seek professional treatment. They prefer over the counter products to reduce the sensitivity when the severity increases.

Hydrodynamic theory by Astron and Brannstorm is accepted most widely out of several theories. According to him the flow of the dentinal fluid was dependent upon the mechanical, thermal, evaporative, and osmotic stimuli. This flow in tubules can activate nerves along the entire canal of the pulp causing pain. Therefore, closing the dentinal tubules is the key approach in the management of dentin hypersensitivity. This can be done possibly by crystal precipitation in the tubule. Various methods and agents are being used for its management for instance laser therapy and fluorine preparations, strontium and zinc chlorides, potassium oxalate and dental adhesives.

Gluma desensitizer is an aqueous solution which contains glutaraldehyde 5% and hydroxyethyl methacrylate (HEMA) 35%. It has been found to be an effective desensitizing agent. It blocks the dentinal tubules intrinsically, countering the mechanism of hydrodynamics that eventually leads to dentin hypersensitivity.

Propolis is a naturally occurring resin. It is brown in colour. It is collected by honey bees from exudates of plants and trees. With the secretions and wax it is modified in the beehives. Honey bees use it to protect their hives and repair any opening or damage.

In homeopathic practices it is widely used as an anti-inflammatory and antiseptic agent. Propolis is composed of resins 50-60%, waxes 30-40%, essential oils 5-10%, pollen 5% and other micro elements like aluminium and calcium.

In dentistry, propolis is found to have multiple clinical uses. It can be used as a mouth freshener in halitosis, as a mouthwash, a relief from denture stomatitis, to heal ulcerations, cervical, dentinal, and root caries sensitivity.

Several studies that were performed in vitro have revealed that, propolis has a significant effect on the reduction of dentin permeability. Studies comparing the desensitizing effect of propolis with gluma desensitizer in-vivo are found to be very few.

MATERIALS AND METHODS Study design and settings A randomized, single blind clinical trial was conducted in the department of Operative dentistry, Dr. Ishrat ul Ebad Khan Institute of Oral Health Sciences, Karachi.

Selection criteria

Patient inclusion criteria:

* Patients aged 18- 60 years.
* Patients who had at least two teeth with dentin hypersensitivity, non carious cervical lesion.
* Patients exhibiting pain scores of ≥ 2 on visual analogue scale.

Patient exclusion criteria:

* Teeth with fractures or cracks in the cervical areas of the teeth.
* Cervical areas that are involved in extensive fillings, dentures or orthodontics appliances.
* Patients having any psychological disease.
* Patients taking analgesics on daily basis.

Withdrawal criteria Failure to complete follow-up after undergoing initial treatment and giving consent.

Method of collection of data Ethical approval Approval was granted by the Institutional review board of Dow University of Health Sciences.

Informed consent All the study participants were informed in detail about the nature of the research procedure, and a written consent was obtained.

Sample size and technique The sample size calculated was 80 teeth, 40 teeth per group (Group A = Propolis, group B = Gluma) carried out using PASS v.11 to independent sample T test at 95% confidence interval and 80% power of test. Calculation was done on mean SD values 0.6+/-0.58 and 0.31+/-0.459 of propolis and gluma respectively.

The sampling technique used in this study was non probability purposive sampling.

Study duration The experimental period of this study was one month. The desensitizing agents were randomly applied to the dentin hypersensitive teeth.

Application procedure:

* First the affected area was cleaned of any debris or plaque.
* Isolation of the affected tooth was done with the help of cotton rolls.
* Tooth surfaces was dried with cotton pellet.
* 30% ethanolic extract of propolis was applied on the dentin hypersensitive site by using a bonding brush then was allowed to dry for 60 seconds.
* Gluma desensitizer was applied according to the manufacturer's instructions.
* Care was taken that the desensitizing agents do not touch any other surface of the oral mucosa.
* Instructions were then given to the patient to not to rinse, eat or drink for 30 minutes after the application of the desensitizing agent.
* Further the patient was asked to avoid the usage of any other desensitizing agent during this one month study period.

The evaporative (air blast) sensitivity test was assessed by application of air from a triple air dental syringe for 1-2 second at a distance of 1 cm from the isolated tooth surface, to avoid desiccation of the dentin surface.

Schiff's sensitivity scale, and visual analogue scale were used to assess dentine hypersensitivity on air blast stimuli at baseline, immediate, after one week of application and after one month of application of the desensitizing agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18- 60 years.
* Patients who have at least one tooth of dentin hypersensitivity on right and left side of the mouth, non carious cervical lesion.
* Patients exhibiting pain scores of at least two on visual analogue scale would be included in the study

Exclusion Criteria:

* Teeth with fractures or cracks in the cervical areas of the teeth.
* Cervical areas that are involved in extensive fillings, dentures or orthodontics appliances.
* Patients who have a history of any psychological diseases.
* Patients who use analgesic/anti-inflammatory medicines on daily basis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
treatment of dentin hypersensitivity | baseline reading will be taken on VAS At day 0 then propolis will be applied.
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading on VAS will be taken immediately after application of Propolis on day 0
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading on VAS will be taken after 1 week of application Propolis
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading on VAS will be taken after 1 month of application of Propolis
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | baseline reading will be recorded on Schiff sensitivity score on day 0, then Propolis will be applied
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score on day 0, immediately after application of Propolis
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score 1 week after application of Propolis
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score 1 month after application of Propolis
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | baseline reading will be taken on VAS at day 0, before application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be taken on VAS at day 0, immediately after application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be taken on VAS 1 week after application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be taken on VAS 1 month after application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | baseline reading will be recorded on Schiff sensitivity score on day 0, then Gluma desensitizer will be applied
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score on day 0, immediately after application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score 1 week after application of Gluma desensitizer
  management of dentin hypersensitivity
treatment of dentin hypersensitivity | reading will be recorded on Schiff sensitivity score 1 month after application of Gluma desensitizer
  management of dentin hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Marina Shah, BDS, Principal Investigator — DUHS
Locations (1):
- Marina Shah, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah M, Jat SA, Aziz M. Comparison of the effect of propolis and Gluma desensitizer on the management of dentin hypersensitivity: A randomized controlled trial. J Pak Med Assoc. 2024 May;74(5):843-847. doi: 10.47391/JPMA.9924. PMID 38783427